CLINICAL TRIAL: NCT03484767
Title: A Longitudinal, Exploratory, Natural History Study to Further Characterize and Describe the Signs and Symptoms of Patients With Organic Acidemias
Brief Title: "The MaP Study": Mapping the Patient Journey in MMA and PA
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-3704-P001
Record Dates: First submitted 2018-03-13; First posted 2018-04-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Methylmalonic Acidemia; Propionic Acidemia
Keywords: methylmalonic acidemia; MMA; organic acidemia; mut deficiency; inborn errors of metabolism; mut0; mut-; PA; PCCA; PCCB; propionic acidemia
MeSH Terms: conditions — Methylmalonic acidemia; Propionic Acidemia; Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methylmalonic Acidemia Participants: Individuals with isolated MMA (mut0 and mut-)
- Propionic Acidemia Participants: Individuals with isolated PA

SUMMARY:
Longitudinal, exploratory, natural history study of patients with MMA due to mut deficiency and PA to characterize the changes in blood disease biomarkers over time and the frequency and severity of clinical events related to their disease.

ELIGIBILITY:
Inclusion Criteria:

MMA Only • Patient has a confirmed diagnosis of isolated MMA due to MUT deficiency (mut0 or mut-) based on the following criteria:

* Elevated plasma/serum/DBS or urine methylmalonic acid levels
* Presence of normal serum/plasma vitamin B12 and plasma homocysteine levels
* Confirmed by molecular genetic testing. Genetic testing can be performed after the administration of informed consent if not available, however, molecular genetic results must be confirmed before the second study visit

PA Only

• Patient has a confirmed diagnosis of isolated PA based on the following criteria:

* Elevated plasma/DBS/urine 2-MC and/or 3-HP
* Elevated plasma/serum/DBS propionylcarnitine (C3)
* Confirmed by genetic testing for mutations of the PCCA or PCCB genes. Genetic testing can be performed after the administration of informed consent if not available, however, molecular genetic results must be confirmed before the second study visit

Both MMA and PA

* Patient (and/or legally authorized representative as applicable to local regulations) is willing and able to comply with study-related assessments and activities
* Patient or legally authorized representative is willing and able to provide informed consent and/or assent as mandated by local regulation

Exclusion Criteria:

* Estimated GFR <30 mL/min/1.73m2 based on age appropriate equations or patients who undergo chronic dialysis
* The patient is pregnant or lactating at the time of screening. (Note: Patients who become pregnant during the study may remain in the study) MMA Only
* Patients diagnosed with isolated MMA cblA, cblB, or cblD enzymatic subtypes or methylmalonyl-CoA epimerase deficiency or combined MMA with homocystinuria PA Only
* Patient has a confirmed diagnosis of multiple carboxylase deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of any age with confirmed diagnosis of isolated MMA due to MUT deficiency (mut0 or mut-) or isolated PA
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Change in plasma methylmalonic acid levels (MMA only) | Baseline through 12 months
Frequency of disease related clinical events in enrolled participants (mut0 and mut- MMA patients) | Baseline through 12 months
Changes in plasma 2-MC levels (PA only) | Baseline through 12 months
Changes in plasma 3-HP levels (PA only) | Baseline through 12 months
Frequency of disease related clinical events in enrolled participants (PA patients) | Baseline through 12 months

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - Stanford Health Services, Stanford, California
  - Emory Univeristy, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seattle Children's Hospital, Seattle, Washington
- France (2):
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Hôpital Necker - Enfants Malades, Paris, Paris
- Hospital de Cruces, Barakaldo, Vizcaya, Spain
- United Kingdom (3):
  - Great Ormond Street Hospital, Bloomsbury, Greater London
  - Birmingham Children's Hospital, Birmingham
  - Manchester University Hospitals, Manchester

IPD SHARING:
Plan to Share IPD: No